CLINICAL TRIAL: NCT03835481
Title: Phase II Long-term Extension Study to Assess the Safety, Tolerability, and Efficacy of BI 730357 in Patients With Moderate-to-severe Plaque Psoriasis
Brief Title: A Study to Test How Well Patients With Plaque Psoriasis Tolerate BI 730357 Over a Longer Period and How Effective it is
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to company decision.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1407-0005; 2018-003487-31 (EudraCT Number)
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Results first posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 25 mg BI 730357 (Experimental): 25 mg BI 730357 + placebo under fasted conditions.
  Interventions: Drug: BI 730357; Drug: Placebo to match BI 730357
- 50 mg BI 730357 (Experimental): 50 mg BI 730357 + placebo under fasted conditions.
  Interventions: Drug: BI 730357; Drug: Placebo to match BI 730357
- 100 mg BI 730357 (Experimental): 100 mg BI 730357 + placebo under fasted conditions.
  Interventions: Drug: BI 730357; Drug: Placebo to match BI 730357
- 200 mg BI 730357 (Experimental): 200 mg BI 730357 + placebo under fasted conditions
  Interventions: Drug: BI 730357; Drug: Placebo to match BI 730357
- 400 mg BI 730357 (Experimental): 400 mg BI 730357 + placebo under fasted conditions.
  Interventions: Drug: BI 730357

INTERVENTIONS:
Drug: BI 730357 — Film-coated tablet
Drug: Placebo to match BI 730357 — Film-coated tablet
  Arms: 100 mg BI 730357; 200 mg BI 730357; 25 mg BI 730357; 50 mg BI 730357

SUMMARY:
To assess long-term safety, tolerability, and efficacy of BI 730357 in patients with moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Woman Of Child Bearing Potential (WOCBP) must be ready and able to use highly effective methods of birth control per International Conference on Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly from date of screening until 4 weeks after last treatment in this trial. A list of contraception methods meeting these criteria is provided in the patient information.
* Patients with moderate-to-severe plaque Psoriasis (PsO) who have completed treatment in the preceding trial without early discontinuation, agree to continue treatment in 1407-0005, and

  * for patients entering from Part 1 of trial 1407-0030

    --- achieve a ≥PASI50 response upon completing the trial 1407-0030 Week 24 end-of-treatment visit
  * for patients entering from Part 2 of trial 1407-0030 --- achieve a ≥PASI50 response upon completing the trial 1407-0030 Week 12 end-of-treatment visit or perceived patient improvement, at the discretion of the Investigator
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.

Exclusion Criteria:

* Nonplaque forms of PsO (including guttate, erythrodermic, or pustular), current druginduced PsO (including a new onset or exacerbation of PsO from, e.g., beta blockers, calcium channel blockers, lithium), active ongoing inflammatory diseases (including but not limited to inflammatory bowel disease (IBD)) other than PsO that might confound trial evaluations.
* Previous enrolment in this trial.
* Currently enrolled in another investigational device or drug trial or is receiving other investigational treatment(s) (with the exception of 1407-0030).
* Intake of any restricted medication or any drug considered likely to interfere with the safe conduct of the trial.
* Any plan to receive a live vaccination during the conduct of the trial.
* Patients not expected to comply with the protocol requirements or not expected to complete the trial as scheduled.
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes the patient an unreliable trial participant or unlikely to complete the trial.
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial.
* Any documented active or suspected malignancy, except appropriately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ carcinoma of uterine cervix.
* Relevant chronic or acute infections including human immunodeficiency virus (HIV), viral hepatitis and tuberculosis.
* Evidence of a disease (including known or suspected IBD, cardiovascular disease), or medical finding that in the opinion of the Investigator is clinically significant and would make the study participant unreliable to adhere to the protocol or to complete the trial, compromise the safety of the patient, or compromise the quality of the data.
* Any suicidal ideation, including grade 4 or 5 in the Columbia Suicide Severity Rating Scale (C-SSRS) in the past 12 months (i.e., active suicidal thought with intent but without specific plan), or active suicidal thought with plan and intent in the past.
* Unwillingness to adhere to the rules of UV-light protection
* Ongoing AEs consistent with intolerance of trial medication (including gastric intolerance) from 1407-0030, that in the opinion of the investigator would compromise the safety of the patient.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (15):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Dermatology Research Associates, Los Angeles, California
  - Southern California Dermatology Inc., Santa Ana, California
  - Hamilton Research, Alpharetta, Georgia
  - Advanced Medical Research PC, Sandy Springs, Georgia
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Clinical Research Center of the Carolinas, Charleston, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Menter Dermatology Research Institute, Dallas, Texas
  - Center for Clinical Studies, Houston, Texas
  - Center for Clinical Studies, Webster, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Canada (10):
  - Dr Chih-ho Hong Medical Inc, Surrey, British Columbia
  - Enverus Medical Research, Surrey, British Columbia
  - Dr. Irina Turchin PC Inc., Fredericton, New Brunswick
  - The Guenther Dermatology Research Centre, London, Ontario
  - DermEdge Research Inc., Mississauga, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - K. Papp Clinical Research Inc., Waterloo, Ontario
  - XLR8 Medical Research Inc., Windsor, Ontario
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - TFS Trial Form Support GmbH, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Universitätsklinikum Münster, Münster

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Gooderham MJ, Mrowietz U, Kadus W, Drda K, Gu H, Vangerow H, Flack M, Korell J, Sofen H, Papp KA. Phase II Randomized Trial of BI 730357, an Oral RORgammat Inhibitor, for Moderate-to-Severe Plaque Psoriasis. J Invest Dermatol. 2025 Aug;145(8):1969-1978.e14. doi: 10.1016/j.jid.2024.12.025. Epub 2025 Jan 21. PMID 39848568
- [Derived] Ooi QX, Kristoffersson A, Korell J, Flack M, L Plan E, Weber B. Bounded integer model-based analysis of psoriasis area and severity index in patients with moderate-to-severe plaque psoriasis receiving BI 730357. CPT Pharmacometrics Syst Pharmacol. 2023 Jun;12(6):758-769. doi: 10.1002/psp4.12948. Epub 2023 May 1. PMID 36919398
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicentre, long-term extension trial in patients with moderate-to-severe plaque psoriasis who completed treatment in the preceding trial 1407-0030 (NCT03635099). Patients rolling over from Part 1 of 1407-0030 remained on their blinded BI 730357 dose treatment, until the open label period of 1407-0005 started at Day 1 of week 13 (dose group 25-200 mg). Patients rolling over from Part 2 of 1407-0030 were assigned at visit 1 to receive open label treatment with 400 mg BI 737357.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Only subjects which met all inclusion and none of the exclusion criteria were included in the trial. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 25 mg BI 730357: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 25 milligram (mg) BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily until end of study (period 2) or received an optional up-titration to 200 mg BI 730357.
- 50 mg BI 730357: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 50 milligram (mg) BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open-label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily until end of study (period 2) or received an optional up-titration to 200 mg BI 730357.
- 100 mg BI 730357: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 100 milligram (mg) BI 730357 and 3 film-coated tablet of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were assigned to 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily until end of study (period 2) or received an optional up-titration to 200 mg BI 730357.
- 200 mg BI 730357: Patients entering from part 1 of 1407-0030 were administered 2 film-coated tablets of 100 milligram (mg) BI 730357 and 2 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were assigned to 200 mg BI 730357 open label dose, receiving 2 film-coated tablets of 100 mg BI 730357 orally administered once daily until end of study (period 2).
- 400 mg BI 730357: Patients entering from part 2 of 1407-0030 were administered open label treatment of 4 film-coated tablets of 100 milligram (mg) BI730357 orally once daily (QD) under fed conditions throughout the trial.
Period: Double-blind Period
Arm/Group | 25 mg BI 730357 | 50 mg BI 730357 | 100 mg BI 730357 | 200 mg BI 730357 | 400 mg BI 730357
Started (Enrolled) | 2 | 20 | 16 | 49 | 78
Completed (Completed week 12) | 2 | 18 | 15 | 46 | 37
Not Completed | 0 | 2 | 1 | 3 | 41
Not completed — Other not stated below | 0 | 0 | 0 | 1 | 1
Not completed — Termination of treatment by sponsor | 0 | 0 | 0 | 0 | 35
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 1 | 0
Period: Open Label Period (After Week 12)
Arm/Group | 25 mg BI 730357 | 50 mg BI 730357 | 100 mg BI 730357 | 200 mg BI 730357 | 400 mg BI 730357
Started (Patients assigned to 25 or 50 mg in part 1 were reassigned to 100 mg in the open label period.) | 0 (0 patients started period 2, patients were switched to 100 mg.) | 0 (0 patients started period 2, patients were switched to 100 mg.) | 35 (Combination of Double-blind period dose groups: 25, 50 and 100 mg.) | 46 | 37
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 35 | 46 | 37
Not completed — Termination of treatment by Sponsor | 0 | 0 | 23 | 31 | 35
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 9 | 1
Not completed — Lost to Follow-up | 0 | 0 | 4 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0
Not completed — Covid-19 related, not due to Adverse event | 0 | 0 | 0 | 1 | 0
Not completed — Other not stated above | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All patients who received at least one dose of treatment in the extension trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg BI 730357 | 50 mg BI 730357 | 100 mg BI 730357 | 200 mg BI 730357 | 400 mg BI 730357 | Total
Number analyzed (Participants) | 2 | 20 | 16 | 49 | 78 | 165
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.0 (2.8) | 47.2 (18.3) | 58.1 (13.5) | 49.9 (13.3) | 44.5 (13.3) | 47.7 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 8 | 7 | 12 | 22 | 49
  Male | 2 | 12 | 9 | 37 | 56 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 6 | 2 | 12 | 23 | 44
  Not Hispanic or Latino | 1 | 14 | 14 | 37 | 55 | 121
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 6 | 7 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 1 | 1 | 6 | 12
  White | 1 | 17 | 13 | 42 | 64 | 137
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Number of participants with treatment emergent adverse events (TEAEs). For dose groups 25 mg - 200 mg BI, TEAEs are reported separately for period 1 and period 2.
  Period 1: All patients who started in period 1 are reported by starting dose (25, 50, 100 and 200 mg).
  Period 2: Only patients who participated in period 2 are reported by dose sequence group.
  For dose group 400 mg BI, TEAEs are reported overall (period 1 + period 2). Number of participants with TEAEs is reported.
Time Frame: For part 1 patients in period 1: Up to 117 days. For part 1 patients in period 2: From week 13 onwards, up to 692 days. For part 2 patients (period 1 + 2): Up to 802 days.
Population: Treated Set (TS): All patients who received at least one dose of treatment in the extension trial. For dose groups 25 mg - 200 mg BI, results are reported separately for period 1 and period 2. For dose group 400 mg BI, results are reported overall (period 1 + period 2).
Measure: Count of Participants; unit: Participants
Groups:
- 25 mg BI - 100 mg BI: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 25 mg BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily until end of study (period 2).
- 25 mg BI - 100 mg BI - 200 mg BI: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 25 mg BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily and were up-titrated to 200 mg BI 730357 once daily until end of study (period 2).
- 50 mg BI - 100 mg BI: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 50 mg BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily until end of study (period 2).
- 50 mg BI - 100 mg BI - 200 mg BI: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 50 mg BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily and were up-titrated to 200 mg BI 730357 once daily until end of study (period 2).
- 100 mg BI - 100 mg BI: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 100 mg BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily until end of study (period 2).
- 100 mg BI - 100 mg BI - 200 mg BI: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 100 mg BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily and were up-titrated to 200 mg BI 730357 once daily until end of study (period 2).
- 200 mg BI - 200 mg BI: Patients entering from part 1 of 1407-0030 were administered 2 film-coated tablets of 100 milligram (mg) BI 730357 and 2 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were assigned to the 200 mg BI 730357 open label dose, receiving 2 film-coated tablets of 100 mg BI 730357 orally administered once daily until end of study (period 2).
Arm/Group | 25 mg BI 730357 | 50 mg BI 730357 | 100 mg BI 730357 | 200 mg BI 730357 | 400 mg BI 730357 | 25 mg BI - 100 mg BI | 25 mg BI - 100 mg BI - 200 mg BI | 50 mg BI - 100 mg BI | 50 mg BI - 100 mg BI - 200 mg BI | 100 mg BI - 100 mg BI | 100 mg BI - 100 mg BI - 200 mg BI | 200 mg BI - 200 mg BI
Number analyzed (Participants) | 2 | 20 | 16 | 49 | 78 | 1 | 1 | 5 | 13 | 6 | 9 | 46
Participants | 0 | 6 | 6 | 10 | 14 | 1 | 0 | 3 | 8 | 3 | 6 | 28

2. Secondary Outcome: Number of Participants With Psoriasis Area and Severity Index (PASI)50/PASI75/PASI90/PASI100 Response at Week 24
Description: Number of participants with PASI50/75/90/100 response, where PASI50/75/90/100 is 50%/75%/90%/100% reduction in PASI score.
  The PASI score is an established measure of clinical efficacy for psoriasis medications, which provides a numeric scoring for patients overall psoriasis disease state, ranging from 0 to 72, with a lower score indicating a better outcome. It is a linear combination of percent of surface area of skin that is affected and the severity of erythema, infiltration, and desquamation over four body regions. The endpoint is based on the percent reduction from baseline, summarized as a dichotomous outcome based on achieving over an X% reduction (or PASI X), where X is 50, 75, 90 and 100.
  The percent reduction from baseline is calculated by % PASI reduction from baseline = ((PASI at baseline - PASI at Visit X) / PASI at baseline) *100, at all visits with PASI collected.
Time Frame: At baseline and at week 24.
Population: Treated Set (TS): All patients who received at least one dose of treatment in the extension trial. Results are reported by dose sequence group. Only participants with non-missing results are reported.
Measure: Count of Participants; unit: Participants
Groups:
- 200 mg BI - 200 mg BI: Patients entering from part 1 of 1407-0030 were administered 2 film-coated tablets of 100 milligram (mg) BI 730357 and 2 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 200 mg BI 730357 open label dose, receiving 2 film-coated tablets of 100 mg BI 730357 orally administered once daily until end of study (period 2).
- 400 mg BI - 400 mg BI: Patients entering from part 2 of 1407-0030 were administered open label treatment of 4 film-coated tablets of 100 milligram (mg) BI730357 orally once daily (QD) under fed conditions throughout the trial. Patients in this group are those part 2 patients who have received treatment for more than 12 weeks.
Arm/Group | 25 mg BI - 100 mg BI | 25 mg BI - 100 mg BI - 200 mg BI | 50 mg BI - 100 mg BI | 50 mg BI - 100 mg BI - 200 mg BI | 100 mg BI - 100 mg BI | 100 mg BI - 100 mg BI - 200 mg BI | 200 mg BI - 200 mg BI | 400 mg BI - 400 mg BI
Number analyzed (Participants) | 1 | 1 | 4 | 13 | 6 | 9 | 45 | 16
Participants
  PASI50 | 0 | 1 | 4 | 12 | 2 | 8 | 33 | 9
  PASI75 | 0 | 1 | 3 | 9 | 2 | 3 | 23 | 6
  PASI90 | 0 | 1 | 1 | 4 | 0 | 2 | 10 | 5
  PASI100 | 0 | 1 | 1 | 2 | 0 | 0 | 3 | 2

3. Secondary Outcome: Number of Participants With Static Physician Global Assessment (sPGA) Clear or Almost Clear Response at Week 24
Description: Number of participants with sPGA clear or almost clear response at week 24. The sPGA is a 5 point score based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. The score ranges from 0 - 4, with a lower score indicating a better outcome.
  0= clear (no signs of psoriasis),
  1. almost clear;
  2. mild;
  3. moderate; 4 = severe (e.g. deep dark red coloration).
Time Frame: At week 24.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mg BI - 100 mg BI | 25 mg BI - 100 mg BI - 200 mg BI | 50 mg BI - 100 mg BI | 50 mg BI - 100 mg BI - 200 mg BI | 100 mg BI - 100 mg BI | 100 mg BI - 100 mg BI - 200 mg BI | 200 mg BI - 200 mg BI | 400 mg BI - 400 mg BI
Number analyzed (Participants) | 1 | 1 | 4 | 13 | 6 | 9 | 45 | 16
Participants | 0 | 1 | 2 | 5 | 1 | 3 | 18 | 7

4. Secondary Outcome: Number of Participants With Static Physician Global Assessment (sPGA) Clear Response at Week 24
Description: Number of participants with sPGA clear response at week 24. The sPGA is a 5 point score based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. The score ranges from 0 - 4, with a lower score indicating a better outcome.
  0= clear (No signs of psoriasis),
  1. almost clear;
  2. mild;
  3. moderate; 4 = severe (e.g. deep dark red coloration).
Time Frame: At week 24.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- 25 mg BI - 100 mg BI - 200 mg BI: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 25 mg BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily until end of study (period 2).
- 50 mg BI - 100 mg BI - 200 mg BI: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 50 mg BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily until end of study (period 2).
- 100 mg BI - 100 mg BI - 200 mg BI: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 100 mg BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily until end of study (period 2).
Arm/Group | 25 mg BI - 100 mg BI | 25 mg BI - 100 mg BI - 200 mg BI | 50 mg BI - 100 mg BI | 50 mg BI - 100 mg BI - 200 mg BI | 100 mg BI - 100 mg BI | 100 mg BI - 100 mg BI - 200 mg BI | 200 mg BI - 200 mg BI | 400 mg BI - 400 mg BI
Number analyzed (Participants) | 1 | 1 | 4 | 13 | 6 | 9 | 45 | 16
Participants | 0 | 1 | 1 | 2 | 0 | 0 | 3 | 2

5. Secondary Outcome: Number of Participants With Psoriasis Area and Severity Index (PASI)50/PASI75/PASI90 or PASI100 Response at Any Time and Loss of PASI Response
Description: The time-to-loss analysis of PASI response was not performed because the analysis would not provide any statistically valid estimates of the parameter due to the premature ending of the trial. Instead, the number of participants with PASI50/75/90/100 response at any time and loss of response at the last efficacy assessment is reported.
  PASI50/75/90/100 is 50%/75%/90%/100% reduction in PASI score. PASI score is a measure of clinical efficacy for psoriasis medications, which ranges from 0 to 72, with a lower score indicating a better outcome.
  A patient was a PASI responder if he or she achieved a response at any time from enrollment to 7 days (Residual effect period (REP)) after last dosing date.
  A patient with the event of loss of response was a responder that lost their PASI response at the last efficacy assessment regardless if it was done within 7 days (REP) after the last dosing date or not.
Time Frame: Up to 802 days.
Population: Treated Set (TS): All patients who received at least one dose of treatment in the extension trial. Only participants with non-missing results are reported. Results are reported per starting dose (50, 100, 200 and 400 mg) for patients who participated only in period 1, and per dose-sequence group for patients who participated in period 1 and period 2.
Measure: Number; unit: Participants
Groups:
- 100 mg BI - 100 mg BI - 200 mg BI: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 100 mg BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily until end of study (period 2).
Arm/Group | 50 mg BI 730357 | 100 mg BI 730357 | 200 mg BI 730357 | 400 mg BI 730357 | 25 mg BI - 100 mg BI | 25 mg BI - 100 mg BI - 200 mg BI | 50 mg BI - 100 mg BI | 50 mg BI - 100 mg BI - 200 mg BI | 100 mg BI - 100 mg BI | 100 mg BI - 100 mg BI - 200 mg BI | 200 mg BI - 200 mg BI | 400 mg BI - 400 mg BI
Number analyzed (Participants) | 2 | 1 | 3 | 41 | 1 | 1 | 5 | 13 | 6 | 9 | 46 | 37
Participants
  PASI50 Responders | 0 | 1 | 2 | 23 | 1 | 1 | 5 | 13 | 6 | 9 | 46 | 30
  PASI50 Loss of Response | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 5 | 3 | 11 | 4
  PASI75 Responders | 0 | 1 | 0 | 12 | 1 | 1 | 4 | 12 | 3 | 6 | 32 | 21
  PASI75 Loss of Response | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 12 | 5
  PASI90 Responders | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 5 | 0 | 3 | 21 | 10
  PASI90 Loss of Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 12 | 2
  PASI100 Responders | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 4 | 0 | 1 | 12 | 4
  PASI100 Loss of Response | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 7 | 1

6. Secondary Outcome: Number of Participants With Static Physician's Global Assessment (sPGA) Clear or Almost Clear Response at Any Time and Loss of sPGA Clear or Almost Clear Response
Description: The time-to-loss analysis of PASI response was not performed because the analysis would not provide any statistically valid estimates of the parameter due to the premature ending of the trial. Instead, the number of participants with sPGA clear or almost clear response at any time, and loss of response at the last efficacy assessment is reported.
  The sPGA is based on the physician's assessment of average thickness, erythema and scaling of all psoriatic lesions. It ranges from 0 to 4, with 0=clear (best outcome), 1=almost clear, 2=mild, 3=moderate and 4=severe (worst outcome).
  A patient was an sPGA responder if he or she achieved a response at any time from enrolment to 7 days (residual effect period (REP)) after last dosing date. A patient with the event of loss of response was a responder that lost their sPGA response at the last efficacy assessment regardless if it was done within 7 days (REP) after the last dosing date or not.
Time Frame: Up to 802 days.
Population: as for outcome 5
Measure: Number; unit: Participants
Groups:
- 200 mg BI - 200 mg BI: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 100 mg BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily until end of study (period 2).
Arm/Group | 50 mg BI 730357 | 100 mg BI 730357 | 200 mg BI 730357 | 400 mg BI 730357 | 25 mg BI - 100 mg BI | 25 mg BI - 100 mg BI - 200 mg BI | 50 mg BI - 100 mg BI | 50 mg BI - 100 mg BI - 200 mg BI | 100 mg BI - 100 mg BI | 100 mg BI - 100 mg BI - 200 mg BI | 200 mg BI - 200 mg BI | 400 mg BI - 400 mg BI
Number analyzed (Participants) | 2 | 1 | 3 | 41 | 1 | 1 | 5 | 13 | 6 | 9 | 46 | 37
Participants
  Resonders | 0 | 1 | 0 | 13 | 0 | 1 | 3 | 9 | 3 | 6 | 32 | 17
  Loss of response | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 4 | 3 | 2 | 18 | 3

7. Secondary Outcome: Number of Participants With Static Physician's Global Assessment (sPGA) Clear Response at Any Time and Loss of sPGA Clear Response
Description: The time-to-loss analysis of PASI response was not performed because the analysis would not provide any statistically valid estimates of the parameter due to the premature ending of the trial. Instead, the number of participants with sPGA clear response at any time, and loss of response at the last efficacy assessment is reported.
  The sPGA is based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions. It ranges from 0 to 4, with 0=clear (best outcome), 1=almost clear, 2=mild, 3=moderate and 4=severe (worst outcome).
  A patient was a sPGA responder if he or she achieved a response at any time from enrolment to 7 days (residual effect period (REP)) after last dosing date.
  A patient with the event of loss of response was a responder that lost their sPGA response at the last efficacy assessment regardless if it was done within 7 days (REP) after the last dosing date or not.
Time Frame: Up to 802 days.
Population: as for outcome 5
Measure: Number; unit: Participants
Groups:
- 50 mg BI - 100 mg BI - 200 mg: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 50 mg BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily until end of study (period 2).
- 100 mg BI - 100 mg - 200 mg BI; 200 mg BI - 200 mg BI: Patients entering from part 1 of 1407-0030 were administered 1 film-coated tablet of 100 mg BI 730357 and 3 film-coated tablets of placebo orally once daily (q.d.) under fasted conditions for the initial 12 week double-blind treatment period (period 1). At day 1 of week 13 (visit 2) patients were reassigned to the 100 mg BI 730357 open label dose, receiving 1 film-coated tablet of 100 mg BI 730357 orally administered once daily until end of study (period 2).
Arm/Group | 50 mg BI 730357 | 100 mg BI 730357 | 200 mg BI 730357 | 400 mg BI 730357 | 25 mg BI - 100 mg BI | 25 mg BI - 100 mg BI - 200 mg BI | 50 mg BI - 100 mg BI | 50 mg BI - 100 mg BI - 200 mg | 100 mg BI - 100 mg BI | 100 mg BI - 100 mg - 200 mg BI | 200 mg BI - 200 mg BI | 400 mg BI - 400 mg BI
Number analyzed (Participants) | 2 | 1 | 3 | 41 | 1 | 1 | 5 | 13 | 6 | 9 | 46 | 37
Participants
  Resonders | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 4 | 0 | 1 | 12 | 4
  Loss of response | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 7 | 1

ADVERSE EVENTS:
Time Frame: From start of treatment until last dose, plus 7 days of residual effect period, up to 802 days.
Description: Treated Set (TS): All participants who received at least one dose of treatment in the extension trial. Arms are not mutually exclusive.
Groups:
- 25 mg BI 730357 (Actual Dose): Patients received 25 mg of BI 730357 orally once daily under fasted conditions in period 1. This group includes all subjects who actually received 25 mg BI 730357.
- 50 mg BI 730357 (Actual Dose): Patients received 50 mg of BI 730357 orally once daily under fasted conditions in period 1. This group includes all subjects who actually received 50 mg BI 730357.
- 100 mg BI 730357 BI (Actual Dose): Patients who received 100 mg of BI 730357 orally once daily under fasted conditions in period 1 and/or period 2. This group includes all subjects who actually received 100 mg BI 730357.
- 200 mg BI 730357 (Actual Dose): Patients received 200 mg of BI 730357 orally once daily under fasted conditions in period 1 and/or period 2. This group includes all subjects who actually received 200 mg BI 730357.
- 400 mg BI 730357 (Actual Dose): Patients received 400 mg of BI 730357 orally once daily under fed conditions throughout the trial. This group includes all subjects who actually received 400 mg BI 730357.
Arm/Group | 25 mg BI 730357 (Actual Dose) | 50 mg BI 730357 (Actual Dose) | 100 mg BI 730357 BI (Actual Dose) | 200 mg BI 730357 (Actual Dose) | 400 mg BI 730357 (Actual Dose)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/20 | 0/36 | 0/72 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/20 | 3/36 | 3/72 | 0/78
Other Adverse Events (participants affected / at risk) | 0/2 | 3/20 | 11/36 | 15/72 | 1/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 25 mg BI 730357 (Actual Dose) (N=2) | 50 mg BI 730357 (Actual Dose) (N=20) | 100 mg BI 730357 BI (Actual Dose) (N=36) | 200 mg BI 730357 (Actual Dose) (N=72) | 400 mg BI 730357 (Actual Dose) (N=78)
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 25 mg BI 730357 (Actual Dose) (N=2) | 50 mg BI 730357 (Actual Dose) (N=20) | 100 mg BI 730357 BI (Actual Dose) (N=36) | 200 mg BI 730357 (Actual Dose) (N=72) | 400 mg BI 730357 (Actual Dose) (N=78)
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 3 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 0
Headache (Nervous system disorders) | 0 | 0 | 3 | 3 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 0

LIMITATIONS AND CAVEATS:
The trial was ended prematurely by the sponsor. As a consequence, primary and secondary endpoints were limited to descriptive outcome measures. The recruitment was completed as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-10-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT03835481/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/81/NCT03835481/SAP_001.pdf